CLINICAL TRIAL: NCT05405387
Title: A Randomized Phase 2 Trial Investigating the Impact of Budesonide Prophylaxis on Incidence of ≥ Grade 2 Diarrhea in Multiple Myeloma (MM) Patients Undergoing Autologous Stem Cell Transplant
Brief Title: Impact of Budesonide on Incidence of ≥ Gr2 Diarrhea in Multiple Myeloma (MM) Patients Undergoing Autologous Stem Cell Transplant
Acronym: IMPACT
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMC Finding
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCI152269
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Plasma Cell Leukemia
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell | interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: Stage one is open-label safety run-in. Stage 2 is randomized, placebo-controlled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To preserve the blind, only the Investigational Drug Services Pharmacy personnel and Data Safety Monitoring Committee (DSMC) at Huntsman Cancer Institute will know treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Run-In Phase (Experimental): Budesonide EC 3 mg three times a day, oral
  Interventions: Drug: Budesonide EC
- Arm 1: Treatment (Experimental): Budesonide EC 3 mg three times a day, oral
  Interventions: Drug: Budesonide EC
- Arm 2: Placebo (Placebo Comparator): Placebo 3 mg three times a day, oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide EC — Subjects will take 3mg of Budesonide or placebo. Dosing will begin on day prior to cell infusion and continue until Day 14 post transplant. Budesonide or placebo will be in capsule formulation. Budesonide or Placebo will be administered orally three times daily (every 8 hours ± 1 hours) with or without food.
  Other Names: Entocort EC
  Arms: Arm 1: Treatment; Run-In Phase
Drug: Placebo — Subjects will take 3mg of Budesonide or placebo. Dosing will begin on day prior to cell infusion and continue until Day 14 post transplant. Budesonide or placebo will be in capsule formulation. Budesonide or Placebo will be administered orally three times daily (every 8 hours ± 1 hours) with or without food.
  Arms: Arm 2: Placebo

SUMMARY:
A randomized placebo controlled, phase 2 study of budesonide in subjects with multiple myeloma undergoing autologous stem cell transplant (ACST). The study includes a run-in period with 20 patients.

DETAILED DESCRIPTION:
The trial will initiate with a safety run-in of 20 pts with a ≥ 5 pts failing to engraft (or having a Grade 4 or higher infection rate) within 18 days as the flag for a potential safety signal.

After all 20 of the patients in the safety run-in have completed follow-up for delayed engraftment (18 days), if the trial is not stopped for a safety signal, then the trial will proceed to a randomized stage. 50 patients will be randomized to placebo and 50 patients will be randomized to budesonide.

Patients in both arms will report toxicities by responding to items from the Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE.) PRO-CTCAE is a patient-reported outcome (PRO) measurement system used to evaluate symptomatic toxicity in patients on cancer clinical trials based on symptom frequency, severity, interference, amount, and presence/absence. PRO-CTCAE responses are scored from 0 (absent) to 4 (very frequent, severe, etc.), or 0/1 for absent/present.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged ≥ 18 years.
* History of histologically confirmed multiple myeloma and/or Plasma Cell Leukemia diagnosis undergoing ASCT who are determined to be fit by the investigator to undergo ASCT with melphalan 200 mg/m2 or melphalan 140 mg/m2 as conditioning.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Adequate organ function as defined as:

  --Hepatic:
  * Total Bilirubin ≤ 2 x institutional upper limit of normal (ULN).
  * AST(SGOT)/ALT(SGPT) ≤ 5 × institutional ULN
* For female subjects who have not undergone surgical sterilization: Negative pregnancy test or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or
    * Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago; or
    * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).

Inclusion Criteria required for Patients Enrolling in Safety Run-In Cohort only:

-Patient must have at least 2.5 x 106 CD34 cells in reserve for use if engraftment is delayed

Exclusion Criteria:

* Ongoing or current use of oral budesonide at the time of enrollment.
* Receiving other investigational agents, unless deemed acceptable after consultation with the PI
* Subjects with moderate or severe pre-existing hepatic impairment as classified according to the Child-Pugh system.
* Prior history or current diagnosis of inflammatory bowel disease, microscopic colitis at baseline.
* Prior history of receiving an allogenic stem cell transplant
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.
* Known prior severe hypersensitivity to melphalan or budesonide or any component in their formulations or compounds of similar composition (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in Section 6.6.1. A washout period of prohibited medications for a period of at least five half-lives or 14 days (whichever is shorter) should occur before the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-05-19 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with delayed engraftment (engraftment after day 18) and severe infection related complications (≥ Grade 4 NCI CTCAE v5). | 18 days
  impact of budesonide prophylaxis on transplant related outcomes in patients with multiple myeloma undergoing ASCT
incidence of Grade 2 or higher diarrhea from the time of ASCT until day 14 post ASCT as measured by NCI Common-Terminology Criteria (CTCAE). | 14 days
  impact of budesonide prophylaxis plus standard of care (SOC) versus standard of care (SOC) alone on the incidence of ≥ Grade 2 diarrhea (NCI CTCAE v5) in multiple myeloma patients receiving high-dose melphalan in preparation for ASCT

SECONDARY OUTCOMES:
proportion of patients reporting "frequent" or "almost constant" diarrhea on Day -1 of transplant on the PRO-CTCAE score | Day -1
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing diarrhea as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
proportion of patients reporting "frequent" or "almost constant" diarrhea on Day 7 of transplant on the PRO-CTCAE score | Day 7
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing diarrhea as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
proportion of patients reporting "frequent" or "almost constant" diarrhea on Day 14 of transplant on the PRO-CTCAE score | Day 14
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing diarrhea as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
proportion of patients reporting "frequent" or "almost constant" diarrhea on Day 30 of transplant on the PRO-CTCAE score | Day 30
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing diarrhea as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
proportion of patients reporting "frequent" or "almost constant" diarrhea 3 months post ACST on the PRO-CTCAE score | 3 Months
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing diarrhea as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
proportion of patients in each arm reporting "frequent" or "almost constant" abdominal pain on Day -1 of transplant on the PRO-CTCAE score | Day -1
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
proportion of patients in each arm reporting "frequent" or "almost constant" abdominal pain on Day 7 aof transplant on the PRO-CTCAE score | Day 7
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
proportion of patients in each arm reporting "frequent" or "almost constant" abdominal pain on Day 14 of transplant on the PRO-CTCAE score | Day 14
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
proportion of patients in each arm reporting "frequent" or "almost constant" abdominal pain on Day 30 of transplant on the PRO-CTCAE score | Day 30
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
proportion of patients in each arm reporting "frequent" or "almost constant" abdominal pain 3 months post ACST on the PRO-CTCAE score | 3 months
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
proportion of patients in each arm reporting "frequent" or "almost constant" nausea on Day 1 of transplant on the PRO-CTCAE score | Day -1
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
proportion of patients in each arm reporting "frequent" or "almost constant" nausea on Day 7 of transplant on the PRO-CTCAE score | Day 7
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
proportion of patients in each arm reporting "frequent" or "almost constant" nausea on Day 14 of transplant on the PRO-CTCAE score | Day 14
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
The proportion of patients in each arm reporting "frequent" or "almost constant" nausea on Day 30 of transplant on the PRO-CTCAE score. | Day 30
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
The proportion of patients in each arm reporting "frequent" or "almost constant" nausea 3 months post ACST on the PRO-CTCAE score. | 3 months
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
The proportion of patients in each arm reporting "frequent" or "almost constant" vomiting on Day 1 of transplant on the PRO-CTCAE score. | Day -1
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
The proportion of patients in each arm reporting "frequent" or "almost constant" vomiting on Day 7 of transplant on the PRO-CTCAE score. | Day 7
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
The proportion of patients in each arm reporting "frequent" or "almost constant" vomiting on Day 14 of transplant on the PRO-CTCAE score. | Day 14
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
The proportion of patients in each arm reporting "frequent" or "almost constant" vomiting on Day 30 of transplant on the PRO-CTCAE score. | Day 30
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
The proportion of patients in each arm reporting "frequent" or "almost constant" vomiting 3 months post ACST on the PRO-CTCAE score. | 3 months
  To demonstrate the superiority of prophylactic budesonide plus standard of care compared to standard of care in reducing alternative gastrointestinal (GI) toxicities (e.g. abdominal pain, nausea) as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (GI domain, fatigue, mouth sore, concentration, and memory)
Length of stay in hospital | up to 30 days
  To assess the effects of prophylactic budesonide plus SOC compared to SOC
Time to engraftment | up to 30 days
  To assess the effects of prophylactic budesonide plus SOC compared to SOC
Proportion of patients using supportive anti-diarrheal and pain medications | up to 30 days
  To assess the effects of prophylactic budesonide plus SOC compared to SOC
Change in Bristol Stool Scale | up to 30 days
  To assess the effects of prophylactic budesonide plus SOC compared to SOC. Scale range is Type 1 to Type 7. A normal stool should be a type 3 or 4, and depending on the normal bowel habits of the individual, should be passed once every one to three days. Type 1 has spent the longest time in the bowel and type 7 the least time.
Incidence of post ASCT infection prior to engraftment | up to 30 days
  To assess the effects of prophylactic budesonide plus SOC compared to SOC
Median score of EORTC QLQ-C30 for participants in each arm | 6 weeks
  To assess the effects of prophylactic budesonide plus SOC compared to SOC
proportion of patients with engraftment syndrome | up to 30 days
  To assess the impact of budesonide prophylaxis on engraftment syndrome in patients with multiple myeloma undergoing ASCT.
Proportion of patients reporting none, mild, moderate, severe or very severe mouth sores as measured by PRO-CTCAE on Day -1 | Day -1
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe mouth sores as measured by PRO-CTCAE on Day 7 | Day 7
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe mouth sores as measured by PRO-CTCAE on Day 14 | Day 14
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe mouth sores as measured by PRO-CTCAE on Day 30 | Day 30
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe mouth sores as measured by PRO-CTCAE 3 months post ACST | 3 months
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very mouth interference with daily activity as a result of their mouth sores as measured by PRO-CTCAE on Day -1 | Day -1
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very mouth interference with daily activity as a result of their mouth sores as measured by PRO-CTCAE on Day 7 | Day 7
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very mouth interference with daily activity as a result of their mouth sores as measured by PRO-CTCAE on Day 14 | Day 14
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very mouth interference with daily activity as a result of their mouth sores as measured by PRO-CTCAE on Day 30 | Day 30
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very mouth interference with daily activity as a result of their mouth sores as measured by PRO-CTCAE 3 months post ACST | 3 months
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe problems with concentration as measured by PRO-CTCAE on Day -1 | Day -1
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe problems with concentration as measured by PRO-CTCAE on Day 7 | Day 7
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe problems with concentration as measured by PRO-CTCAE on Day 14 | Day 14
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe problems with concentration as measured by PRO-CTCAE on Day 30 | Day 30
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe problems with concentration as measured by PRO-CTCAE 3 months post ACST | 3 months
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of concentration problems as measured by PRO-CTCAE on Day -1 | Day -1
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of concentration problems as measured by PRO-CTCAE on Day 7 | Day 7
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of concentration problems as measured by PRO-CTCAE on Day 14 | Day 14
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of concentration problems as measured by PRO-CTCAE on Day 30 | Day 30
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of concentration problems as measured by PRO-CTCAE 3 months post ACST | 3 months
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe problems with memory as measured by PRO-CTCAE on Day -1 | Day -1
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe problems with memory as measured by PRO-CTCAE on Day 7 | Day 7
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe problems with memory as measured by PRO-CTCAE on Day 14 | Day 14
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe problems with memory as measured by PRO-CTCAE on Day 30 | Day 30
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe problems with memory as measured by PRO-CTCAE 3 months post ACST | 3 months
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of problems with memory as measured by PRO-CTCAE on Day -1 | Day -1
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of problems with memory as measured by PRO-CTCAE on Day 7 | Day 7
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of problems with memory as measured by PRO-CTCAE on Day 14 | Day 14
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of problems with memory as measured by PRO-CTCAE on Day 30 | Day 30
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of problems with memory as measured by PRO-CTCAE 3 months post ACST | 3 months
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe fatigue as measured by PRO-CTCAE on Day -1 | Day -1
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe fatigue as measured by PRO-CTCAE on Day 7 | Day 7
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe fatigue as measured by PRO-CTCAE on Day 14 | Day 14
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe fatigue as measured by PRO-CTCAE on Day 30 | Day 30
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, mild, moderate, severe or very severe fatigue as measured by PRO-CTCAE 3 months post ACST | 3 months
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of fatigue as measured by PRO-CTCAE on Day -1 | Day -1
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of fatigue as measured by PRO-CTCAE on Day 7 | Day 7
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of fatigue as measured by PRO-CTCAE on Day 14 | Day 14
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of fatigue as measured by PRO-CTCAE on Day 30 | Day 30
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)
Proportion of patients reporting none, a little bit, somewhat, quite a bit or very much interference with daily activity as a result of fatigue as measured by PRO-CTCAE 3 months post ACST | 3 months
  descriptively assess in both the prophylactic budesonide arm and the standard of care arms the following toxicities as measured by Patient-Reported Outcome Common Terminology Criteria (PRO-CTCAE) (fatigue, mouth sores, concentration, and memory)

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Rehman Mohy-ud-din, MBBS, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No